CLINICAL TRIAL: NCT03770533
Title: Identifying Patients With Suspicion of Infection in the ED Who Have Low Disease Severity Using Midregional Proadrenomedullin (MR-proADM) - Pilot Study
Brief Title: Identifying Patients With Suspicion of Infection in the ED Who Have Low Disease Severity Using MR-proADM - Pilot Study
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IDEAL pilot
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Patients Presenting With Suspicion of Infection to the ED

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MR-proADM guided (Other)
  Interventions: Other: MR-proADM guided
- Standard Care (No Intervention)

INTERVENTIONS:
Other: MR-proADM guided — MR-proADM value together with routine clinical evaluation identifies patients with a low 14 day mortality risk who do not need to be hospitalized
  Arms: MR-proADM guided

SUMMARY:
Emergency departments (ED) are becoming increasingly over-crowded, with patients facing prolonged waiting times. Therefore, a safe and rapid assessment that identifies patients with low severity that could be treated as outpatients is essential for improving the workflow within the ED.

The rationale of this IDEAL study is to provide guidance to safely decrease the number of hospital admissions through identification of low risk patients with the biomarker MR-proADM. This will be tested in a pilot study first.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting to the ED with suspicion of infection
* Age ≥18 years
* Written Informed Consent obtained

Exclusion Criteria:

* Recent major trauma or surgery
* End stage renal failure requiring dialysis
* Terminal disease and/or very severe medical co-morbidity where death has to be expected in the next 6 months, e.g. due to malignancy, cardiac, renal or hepatic failure
* Patients those source of infection always requires hospital admission or never requires hospital admission.
* Patients who cannot be discharged for other than medical reasons
* Patient participates in any other interventional clinical trial
* Patients with active intravenous drug use
* Pregnant or lactating women
* Patients who are institutionalized by official or judicial order
* Dependents of the sponsor, the CRO, the study site or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients admitted to the hospital | 14 days

SECONDARY OUTCOMES:
28 days all-cause hospital re-admission (corrected for mortality) | 28 days
Number of patients re-presenting to the ED within 28 days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gonzalez del Castillo, Principal Investigator — Hospital Clinico San Carlos
Locations (4):
- Spain (4):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Virgen Macarena, Seville

REFERENCES:
- [Derived] Gonzalez Del Castillo J, Clemente-Callejo C, Llopis F, Irimia A, Oltra-Hostalet F, Rechner C, Schwabe A, Fernandez-Rodriguez V, Sanchez-Mora C, Giol-Amich J, Prieto-Garcia B, Bardes-Robles I, Ortega-de Heredia MD, Garcia-Lamberechts EJ, Navarro-Bustos C; INFURG-SEMES investigators. Midregional proadrenomedullin safely reduces hospitalization in a low severity cohort with infections in the ED: a randomized controlled multi-centre interventional pilot study. Eur J Intern Med. 2021 Jun;88:104-113. doi: 10.1016/j.ejim.2021.03.041. Epub 2021 Apr 24. PMID 33906810